CLINICAL TRIAL: NCT04710576
Title: AGAVE-201, A Phase 2, Open-label, Randomized, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of Axatilimab at 3 Different Doses in Patients With Recurrent or Refractory Active Chronic Graft Versus Host Disease Who Have Received at Least 2 Lines of Systemic Therapy
Brief Title: A Study of Axatilimab at 3 Different Doses in Participants With Chronic Graft Versus Host Disease (cGVHD)
Acronym: AGAVE-201
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-6352-0504; 2024-512978-99-00 (EU CTIS Number)
Record Dates: First submitted 2021-01-05; First posted 2021-01-14 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-01

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: cGVHD; AGAVE-201; GVHD; graft versus host disease; graft-versus-host-disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease | interventions — axatilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Axatilimab Dose Cohort 1 (Experimental): Participants will be administered axatilimab 0.3 milligrams (mg)/kilogram (kg) intravenously (IV) every 2 weeks for up to 2 years.
  Interventions: Drug: Axatilimab
- Axatilimab Dose Cohort 2 (Experimental): Participants will be administered axatilimab 1 mg/kg IV every 2 weeks for up to 2 years.
  Interventions: Drug: Axatilimab
- Axatilimab Dose Cohort 3 (Experimental): Participants will be administered axatilimab 3 mg/kg IV every 4 weeks for up to 2 years.
  Interventions: Drug: Axatilimab

INTERVENTIONS:
Drug: Axatilimab — Axatilimab is a high-affinity antibody targeting the colony stimulating factor 1 receptor (CSF-1R). CSF-1R signaling has been demonstrated in nonclinical studies to be the key regulatory pathway involved in the expansion and infiltration of donor-derived macrophages that mediate the disease processes involved in cGVHD.
  Other Names: Niktimvo; SNDX-6352

SUMMARY:
This is a Phase 2 study to evaluate the efficacy, safety, and tolerability of axatilimab at 3 different dose levels in participants with recurrent or refractory active chronic graft versus host disease (cGVHD) who have received at least 2 prior lines of systemic therapy.

DETAILED DESCRIPTION:
AGAVE-201 is a Phase 2, open-label, randomized, multicenter study to evaluate the efficacy, safety, and tolerability of axatilimab in participants with recurrent or refractory active cGVHD after failure of at least 2 prior lines of systemic therapy due to progression of disease, intolerability, or toxicity.

Participants will be randomized to receive 1 of 3 different axatilimab treatment regimens in 28-day treatment cycles for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 2 years of age or older, at the time of signing the informed consent.
2. Participants who are allogeneic hematopoietic stem cell transplantation (HSCT) recipients with active cGVHD requiring systemic immune suppression. Active cGVHD is defined as the presence of signs and symptoms of cGVHD per 2014 NIH Consensus Development Project on Criteria for Clinical trials in cGVHD.
3. Participants with refractory or recurrent active cGVHD despite at least 2 lines of systemic therapy.

   * Refractory disease defined as meeting any of the following criteria:

     * The development of 1 or more new sites of disease while being treated for cGVHD.
     * Progression of existing sites of disease despite at least 1 month of standard or investigation therapy for cGVHD.
     * Participants who have not achieved a response within 3 months on their prior therapy for cGVHD and for whom the treating physician believes a new systemic therapy is required.
   * Recurrent cGVHD is active, symptomatic disease (after an initial response to prior therapy) as defined, based on the NIH 2014 consensus criteria, by organ-specific or global assessment or for which the physician believes that a new line of systemic therapy is required.
4. Participants may have persistent, active acute and cGVHD manifestations (overlap syndrome), as defined by 2014 NIH Consensus Development Project on Criteria for Clinical trials in cGVHD.
5. Karnofsky Performance Scale of ≥60 (if aged 16 years or older); Lansky Performance Score of ≥60 (if aged <16 years)
6. Adequate organ and bone marrow functions evaluated during the 14 days prior to randomization.
7. Creatinine clearance (CrCl) ≥30 milliliter/minute based on the Cockcroft-Gault formula in adult participants and Schwartz formula in pediatric participants.
8. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
9. Concomitant use a of systemic corticosteroid is allowed but not required. Topical and inhaled corticosteroid agents are allowed. If a participant is taking corticosteroids at study randomization, they must be on a stable dose of corticosteroids for at least 2 weeks prior to Cycle 1 Day 1.
10. Concomitant use of CNI or mammalian target of repamycin (mTOR) inhibitors (sirolimus or everolimus) is allowed but not required.
11. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol. A parent/guardian should provide consent for pediatric participants unable to provide consent themselves; in addition, where applicable pediatric participants should sign their own assent form.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has acute GVHD without manifestations of cGVHD.
2. Any evidence (histologic, cytogenetic, molecular, hematologic, or mixed) of relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening.
3. History of acute or chronic pancreatitis.
4. History of myositis.
5. History or other evidence of severe illness, uncontrolled infection or any other conditions that would make the participant, in the opinion of the Investigator, unsuitable for the study.
6. Participants with acquired immune deficiency syndrome (AIDS).
7. Hepatitis B (defined as hepatitis B virus [HBV] surface antigen positive and HBV core antibody positive, with positive HBV deoxyribonucleic acid [DNA], or HBV positive core antibody alone with positive HBV DNA. Hepatitis C (defined as positive hepatitis C [HCV] antibody with positive HCV ribonucleic acid [RNA]).
8. Diagnosed with another malignancy (other than malignancy for which transplant was performed) within 3 years of randomization, unless previously treated with curative intent and approved by Sponsor's Medical Monitor (for example, completely resected basal cell or squamous cell carcinoma of the skin, resected in situ cervical malignancy, resected breast ductal carcinoma in situ, or low-risk prostate cancer after curative resection).
9. Female participant who is pregnant or breastfeeding.
10. Previous exposure to CSF1-R targeted therapies.
11. Taking agents for treatment of cGVHD other than corticosteroids or either a CNI or mTOR inhibitor is prohibited.
12. For approved or commonly used agents, other than corticosteroids, CNI and mTOR inhibitor, a washout of 2 weeks or 5 half-lives, whichever is shorter, is required at study enrollment.
13. Receiving another investigational treatment within 28 days of randomization.
14. Participants should not be participating in any other interventional study. Pediatric participants are encouraged to also participate in the ongoing developmental studies of the Pediatric cGVHD Symptom Scale (PCSS).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vedran Radojcic, M.D., Study Director — Syndax Pharmaceuticals
Locations (120):
- United States (47):
  - University of Alabama at Birmingham - Children's of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida (UF), Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Weill Medical College of Cornell University, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Forest, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Cleveland Clinic Foundation, Lyndhurst, Ohio
  - University of Oklahoma - Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Intermountain Healthcare, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - The Royal Children's Hospital, Parkville, Victoria
  - Westmead Hospital, Westmead
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven, Leuven
  - AZ Delta, Roeselare
- Canada (4):
  - Vancouver Coastal Health Authority, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Center - Research Institute, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
- France (11):
  - CHU de Grenoble, La Tronche, Auvergne-Rhône-Alpes
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg, Grand Est
  - IUCT-Oncopole, Toulouse, Haure-Garrone
  - CHU Amiens Picardie - Hopital Sud, Amiens, Hauts-de-France
  - CHRU de Lille - Hopital Claude Huriez, Lille, Hauts-de-France
  - CHRU de Nancy - Hôpitaux de Brabois, Nancy
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Hopital Pitie Salpetriere, Paris
  - CHU Bordeaux - Hopital Haut-Leveque - Centre François Magendie, Pessac
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (6):
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsmedizin der Johannes Gutenberg - Universitaet Mainz, Mainz
  - Universitaetsklinikum Muenster, Münster
  - Universitatsklinikum Regensburg, Regensburg
- Greece (3):
  - General Hospital of Thessaloniki G. Papanikolaou - Hematology Department, BMT Unit, Eksochi, Thessaloniki
  - University Hospital of West Attica - Attikon - Hematology Division, Athens
  - University General Hospital of Patras, Pátrai
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center Ein Karem, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - ASST di Monza-Ospedale San Gerardo, Monza
  - Fondazione Monza e Brianza per il Bambino e la sua Mamma, Monza
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinica Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
  - AOU Citta della Salute e della Scienza di Torino - Ospedale Regina Margherita, Torino
  - Citta della Salute e della Scienza di Torino - Ospedale le Molinette, Torino
- Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Oddzial w Gliwicach - Klinika Transplantacji Szpiku i Onkohematologii, Gliwice, Poland
- Portugal (2):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, E.P.E. (IPO-Lisboa), Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- Singapore (3):
  - National University Hospital, Singapore
  - KK Women's and Children hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (4):
  - Pusan National University Hospital, Busan
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (13):
  - Hospital Universitario Virgen del Rocio, Seville, Seville
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Complejo Hospitalario Universitario de Granada - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marquis de Valdecilla, Santander
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (6):
  - Bristol Royal Hospital for Children, Bristol
  - University Hospital of Wales, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - Hammersmith Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - Royal Marsden Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolff D, Cutler C, Lee SJ, Pusic I, Bittencourt H, White J, Hamadani M, Arai S, Salhotra A, Perez-Simon JA, Alousi A, Choe H, Kwon M, Bermudez A, Kim I, Socie G, Chhabra S, Radojcic V, O'Toole T, Tian C, Ordentlich P, DeFilipp Z, Kitko CL; AGAVE-201 Investigators. Axatilimab in Recurrent or Refractory Chronic Graft-versus-Host Disease. N Engl J Med. 2024 Sep 19;391(11):1002-1014. doi: 10.1056/NEJMoa2401537. PMID 39292927

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The primary analysis results are reported. The final results will be posted after completion of the study.
Groups:
- Axatilimab 0.3 mg/kg Q2W: Participants received axatilimab 0.3 milligrams (mg)/kilogram (kg) intravenously (IV) every 2 weeks (Q2W) (Days 1 and 15 of each 4-week cycle) for up to 2 years.
- Axatilimab 1 mg/kg Q2W: Participants received axatilimab 1 mg/kg IV Q2W (Days 1 and 15 of each 4-week cycle) for up to 2 years.
- Axatilimab 3 mg/kg Q4W: Participants received axatilimab 3 mg/kg IV every 4 weeks (Q4W) (Day 1 of each 4-week cycle) for up to 2 years.
Period: Overall Study
Arm/Group | Axatilimab 0.3 mg/kg Q2W | Axatilimab 1 mg/kg Q2W | Axatilimab 3 mg/kg Q4W
Started | 80 | 81 | 80
Received at Least 1 Dose of Study Drug | 79 | 81 | 79
Completed | 0 | 1 | 1
Not Completed | 80 | 80 | 79
Not completed — Participants still in the study | 73 | 70 | 60
Not completed — Death | 2 | 7 | 12
Not completed — Withdrawal by Subject | 4 | 3 | 7
Not completed — Sponsor decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set for each dose level included all participants randomized to the dose level.
Groups:
- Axatilimab 0.3 mg/kg Q2W: Participants received axatilimab 0.3 mg/kg IV Q2W (Days 1 and 15 of each 4-week cycle) for up to 2 years.
- Axatilimab 3 mg/kg Q4W: Participants received axatilimab 3 mg/kg IV Q4W (Day 1 of each 4-week cycle) for up to 2 years.
- Total: Total of all reporting groups
Arm/Group | Axatilimab 0.3 mg/kg Q2W | Axatilimab 1 mg/kg Q2W | Axatilimab 3 mg/kg Q4W | Total
Number analyzed (Participants) | 80 | 81 | 80 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (16.88) | 54.0 (12.65) | 50.8 (16.02) | 51.4 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 27 | 90
  Male | 47 | 51 | 53 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 5 | 19
  Not Hispanic or Latino | 73 | 69 | 73 | 215
  Unknown or Not Reported | 2 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 4 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 2 | 1 | 5
  White | 68 | 70 | 62 | 200
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in the First 6 Cycles as Defined by the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-Versus-Host Disease (cGVHD)
Description: The ORR was defined as the percentage of participants with objective response (complete response [CR] or partial response [PR]). CR was defined as resolution of all manifestations in each organ or site, and PR was defined as improvement in at least 1 organ or site without progression in any other organ or site.
Time Frame: First 6 cycles (up to Cycle 7 Day 1; each cycle = 4 weeks)
Population: The ITT analysis set for each dose level included all participants randomized to the dose level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axatilimab 0.3 mg/kg Q2W | Axatilimab 1 mg/kg Q2W | Axatilimab 3 mg/kg Q4W
Number analyzed (Participants) | 80 | 81 | 80
percentage of participants | 73.8 [62.7 to 83.0] | 66.7 [55.3 to 76.8] | 50.0 [38.6 to 61.4]

2. Secondary Outcome: ORR on Study as Defined by the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD
Time Frame: Up to 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants With a Clinically Significant Improvement in Normalized Score on the Modified Lee Symptom Scale
Time Frame: Up to 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from initial partial response or complete response until documented progression of cGVHD, start of new therapy, or death for any reason.
Time Frame: Up to 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Sustained Response Rate
Description: Sustained response rate is defined as the number of participants with objective response lasting for at least 20 weeks (140 days) from the time of initial response. Responses will be assessed based on the 2014 NIH Consensus Development Project on Clinical Trials in cGVHD.
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Organ-specific Response Rate
Description: Organ-specific response is defined as the number of participants with objective response for the nine individual organs based on 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD (skin, eyes, mouth, esophagus, upper gastrointestinal [GI], lower GI, liver, lungs and joints and fascia).
Time Frame: Up to 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Joints and Fascia Response Rate Based on Refined NIH Response Algorithm for cGVHD
Time Frame: Up to 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Percent Reductions in Average Daily Doses (or Equivalent) of Corticosteroid
Time Frame: Up to 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Number of Participants Who Discontinue Corticosteroid Use
Time Frame: Up to 2 years
Reporting Status: Not Posted

10. Secondary Outcome: Percent Reductions in Average Daily Doses (or Equivalent) of Calcineurin Inhibitors (CNI)
Time Frame: Up to 2 years
Reporting Status: Not Posted

11. Secondary Outcome: Number of Participants Who Discontinue CNIs
Time Frame: Up to 2 years
Reporting Status: Not Posted

12. Secondary Outcome: Change From Baseline in Circulating Monocyte Number and Phenotype (CD14/16)
Time Frame: Baseline, up to 2 years
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants With Anti-Drug Antibody
Time Frame: Up to 2 years
Reporting Status: Not Posted

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to Time of Last Measurable Concentration (AUC0-t)
Time Frame: Approximately 12 months
Reporting Status: Not Posted

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Time Frame: Up to 2 years
Reporting Status: Not Posted

16. Secondary Outcome: Change From Baseline in Bone Turnover Markers
Time Frame: Baseline, up to 2 years
Reporting Status: Not Posted

17. Secondary Outcome: Change From Baseline in Bone Density
Time Frame: Baseline, up to 2 years
Reporting Status: Not Posted

18. Secondary Outcome: Change From Baseline in Colony Stimulating Factor 1 (CSF-1) and Interleukin 34 (IL-34) Levels
Time Frame: Baseline, up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 2 years
Description: As pre-specified, All-cause mortality data were collected and reported for all enrolled participants; and Serious and Non-serious adverse events data were collected and reported for all participants who received at least 1 dose of study drug during the study.
Arm/Group | Axatilimab 0.3 mg/kg Q2W | Axatilimab 1 mg/kg Q2W | Axatilimab 3 mg/kg Q4W
All-Cause Mortality (participants affected / at risk) | 2/80 | 7/81 | 12/80
Serious Adverse Events (participants affected / at risk) | 30/79 | 33/81 | 38/79
Other Adverse Events (participants affected / at risk) | 74/79 | 78/81 | 78/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axatilimab 0.3 mg/kg Q2W (N=79) | Axatilimab 1 mg/kg Q2W (N=81) | Axatilimab 3 mg/kg Q4W (N=79)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 1
Acute graft versus host disease (Immune system disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Chronic graft versus host disease (Immune system disorders) | 1 | 0 | 0
Overlap syndrome (Immune system disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 2 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 2 | 0
COVID-19 (Infections and infestations) | 2 | 4 | 5
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 2
Campylobacter infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 3 | 3
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 0
Cryptosporidiosis infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 1 | 0 | 0
Enterovirus infection (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis astroviral (Infections and infestations) | 1 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 2 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 1
Meningitis enteroviral (Infections and infestations) | 0 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 1 | 0
Mycobacterial infection (Infections and infestations) | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1
Oral infection (Infections and infestations) | 0 | 1 | 0
Parainfluenzae viral bronchitis (Infections and infestations) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 8 | 4
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1
Pseudomonal skin infection (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 2 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Superinfection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0
Sapovirus test positive (Investigations) | 1 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axatilimab 0.3 mg/kg Q2W (N=79) | Axatilimab 1 mg/kg Q2W (N=81) | Axatilimab 3 mg/kg Q4W (N=79)
Anaemia (Blood and lymphatic system disorders) | 10 | 6 | 10
Tachycardia (Cardiac disorders) | 5 | 0 | 2
Dry eye (Eye disorders) | 4 | 2 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 4
Periorbital oedema (Eye disorders) | 2 | 19 | 23
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 3 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 13 | 18 | 7
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 5 | 6 | 1
Nausea (Gastrointestinal disorders) | 13 | 14 | 7
Vomiting (Gastrointestinal disorders) | 5 | 4 | 8
Chills (General disorders) | 5 | 5 | 3
Face oedema (General disorders) | 0 | 3 | 7
Fatigue (General disorders) | 18 | 16 | 21
Influenza like illness (General disorders) | 5 | 3 | 3
Non-cardiac chest pain (General disorders) | 4 | 4 | 0
Oedema peripheral (General disorders) | 7 | 12 | 8
Pyrexia (General disorders) | 9 | 9 | 8
Bronchitis (Infections and infestations) | 6 | 3 | 0
COVID-19 (Infections and infestations) | 12 | 14 | 6
Influenza (Infections and infestations) | 4 | 3 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3 | 7
Pneumonia (Infections and infestations) | 2 | 5 | 4
Respiratory syncytial virus infection (Infections and infestations) | 5 | 0 | 3
Respiratory tract infection (Infections and infestations) | 4 | 3 | 1
Rhinovirus infection (Infections and infestations) | 2 | 2 | 4
Sinusitis (Infections and infestations) | 5 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 13 | 11 | 8
Viral upper respiratory tract infection (Infections and infestations) | 1 | 5 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 5 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 3 | 1
Alanine aminotransferase increased (Investigations) | 10 | 18 | 31
Amylase increased (Investigations) | 3 | 10 | 34
Aspartate aminotransferase increased (Investigations) | 11 | 31 | 43
Blood alkaline phosphatase increased (Investigations) | 5 | 4 | 17
Blood creatine phosphokinase increased (Investigations) | 9 | 26 | 49
Blood creatinine increased (Investigations) | 5 | 6 | 4
Blood lactate dehydrogenase increased (Investigations) | 11 | 22 | 32
Gamma-glutamyltransferase increased (Investigations) | 8 | 16 | 21
Lipase increased (Investigations) | 9 | 21 | 39
Platelet count decreased (Investigations) | 7 | 3 | 1
SARS-CoV-2 test positive (Investigations) | 4 | 5 | 2
Weight decreased (Investigations) | 2 | 7 | 5
Decreased appetite (Metabolism and nutrition disorders) | 7 | 3 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 8 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 6 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 7 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 6 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 10 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 16 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 6 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 8 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Dizziness (Nervous system disorders) | 8 | 4 | 5
Headache (Nervous system disorders) | 15 | 14 | 16
Dysuria (Renal and urinary disorders) | 4 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 7 | 12
Rash (Skin and subcutaneous tissue disorders) | 5 | 5 | 3
Hypertension (Vascular disorders) | 5 | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the multi-center Study shall not be made before the first multi-site publication by Sponsor or Publications Committee. No Public Presentation by Institution or Investigator will be made until Study Documentation/Results from all sites are received and analyzed by Sponsor. Separate publication by Investigator will be delayed for a period of 18 months until the initial publication by Committee or Sponsor, or a determination is made not to make such publication.

DOCUMENTS (2):
  • Study Protocol (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04710576/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04710576/SAP_001.pdf